CLINICAL TRIAL: NCT05316246
Title: Efficacy and Safety of Brentuximab Vedotin in Combination With Tislelizumab for the Treatment of CD30-positive Relapsed/Refractory NK/T-cell Lymphoma
Brief Title: Efficacy and Safety of BV With Tislelizumab for the Treatment of CD30+ Relapsed/Refractory NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Takeda (Industry); BeiGene (Industry)
Responsible Party: Principal Investigator, Peng Liu, Chief of hematology department, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSXY-NKT-01
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: NK/T Cell Lymphoma Nos
MeSH Terms: interventions — Brentuximab Vedotin; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CD30-positive Relapsed/Refractory NK/T-cell Lymphoma (Experimental): Brentuximab vedotin will be administered as 1.8 mg/kg IV infusion on Day 1 of each 3-week cycle. PD-1 inhibitor tislelizumab will be administered as 200 mg on Day 1 of each 3-week cycle. Patients will receive maximum of 8 cycles if they do not meet the criteria for removal from the study. Patients will be assessed for overall response using the Revised Response Criteria for Malignant Lymphoma (Lugano 2014). Dedicated computed tomography (CT) scans (neck, chest, abdomen, and pelvis) will be performed at Baseline and at Cycles 2, 4 and 8, and positron emission tomography (PET) scans will be performed at Baseline and at Cycles 4 and 8.
  Interventions: Drug: Brentuximab Vedotin in Combination with Tislelizumab

INTERVENTIONS:
Drug: Brentuximab Vedotin in Combination with Tislelizumab — Brentuximab vedotin will be administered after diluted with 100 ml normal saline as an IV infusion over approximately 30 minutes on Day 1 of each 21-day cycle at a dose of 1.8 mg/kg. Tislelizumab will be administered after diluted with 100 ml normal saline as an IV infusion over approximately 30 minutes on Day 1 of each 21-day cycle at a fixed dose of 200 mg. The rationale of fixed dose of Tislelizumab is according to the drug description, which is based on previous I/II phase clinical trial results of Tislelizumab. The time interval between administration of tislelizumab and brentuximab vedotin should be not less than 2 hours, and thereafter, the dosing cycle of tislelizumab is synchronized with that of brentuximab vedotin.

SUMMARY:
This is a single-arm, open-label, multicenter, phase 2 study designed to evaluate the efficacy and safety of brentuximab vedotin combined with PD-1 inhibitor tislelizumab in Chinese patients with relapsed/refractory CD30+ NK/CL. Brentuximab vedotin will be administered as 1.8 mg/kg IV infusion on Day 1 of each 3-week cycle. PD-1 inhibitor tislelizumab will be administered as 200 mg on Day 1 of each 3-week cycle. Patients will receive maximum of 8 cycles if they do not meet the criteria for removal from the study. Patients will be assessed for overall response using the Revised Response Criteria for Malignant Lymphoma (Lugano 2014). Dedicated computed tomography (CT) scans (neck, chest, abdomen, and pelvis) will be performed at Baseline and at Cycles 2, 4 and 8, and positron emission tomography (PET) scans will be performed at Baseline and at Cycles 4 and 8. No additional PET scanning is required beyond Cycle 8 unless clinically indicated (for example, suspected of disease progression). The disease symptoms will be assessed at Baseline and on Day 1 of each cycle. Patients may continue study treatment until the sooner of disease progression, unacceptable toxicity, or completion of 8 cycles. Patients who discontinue study treatment for any reason other than withdrawal of consent will have safety follow-up assessments through 30 days after the last dose of 、study drug (end of treatment [EOT]). Patients who discontinue study treatment with stable disease (SD), responses and progression disease (PD) will be followed for 1-year PFS rate and 1-year OS rate. The CT scan, PET-CT and laboratory examination will be followed based on clinical practice. The study will be closed when all patients enrolled have completed the required follow-up.Toxicity will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0 Laboratory values, vital signs, and electrocardiograms (ECGs) will be obtained to evaluate the safety and tolerability of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18~75 years
* Histopathology and immunohistochemistry confirmed diagnosis of NK/T-cell lymphoma according to WHO 2016 criteria
* ≥10% CD30 positive for tumor tissue immunohistochemistry
* Previously treated with asparaginase-based regimens (refractory or relapsed after initial remission)
* PET/CT or CT/MRI with at least one objectively measurable or evaluable lesion
* ECOG Performance score 0-2
* The laboratory test within 1 week before enrollment meets the following conditions:
* Blood routine: absolute neutrophil count≥1,500/uL, Leukocytes≥3,000/mm3, Hb>8.0g/dL, PLT>100 ×10*9/L. Liver function: ALT, AST≤ 2.5 times the upper limit of normal, TBIL ≤1.5 times the upper limit of normal. Renal function: Cr >2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute , Amylase and/or lipase ≤1.5 x ULN, Coagulation : plasma fibrinogen ≥ 1.0g/L. Cardiac function: LVEF≥50%, ECG does not suggest any acute myocardial infarction, arrhythmia or atrioventricular conduction above I Blocking,
* Sign the informed consent form,
* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time from the time of signing informed consent through six months after the last dose of study drug
* Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months during entire study treatment period and through 6 months after the last dose of study drug,
* Voluntary compliance with research protocols, follow-up plans, laboratory and auxiliary examinations.

Exclusion Criteria:

* Serious active infection requiring ICU treatment.
* Patients with any active viral, bacterial, or fungal infections that require intravenous antibiotics within 2 weeks before the first dose of the study drug
* Known HIV infection or active infection with HBV, HCV. Patients who are infected with HBV but not active hepatitis at the same time are not excluded.
* Serious complications such as fulminant DIC.
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
* Peripheral neuropathy ≥ Grade 2 (NCI-CTCAE version 5.0 ).
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML
* Significant organ dysfunction: such as respiratory failure, NYHA classification Class III or IV, chronic congestive heart failure, decompensation Hepatic or renal insufficiency, high blood pressure and diabetes that cannot be controlled despite active treatment, and cerebral vascular thrombosis or hemorrhagic time within the past 6 months.
* Pregnant and lactating women.
* Had a history of autoimmune diseases, and disease was active in the last 6 months, and was still taking oral immunosuppressant in the past three months, with daily prednisone dose greater than 10 mg
* Patients who are known to be seriously allergic to any of the drugs in the study regimen (e.g. life-threatening allergic symptoms such as anaphylactic shock).
* Patients combined with other tumors who require surgery or chemotherapy within 6 months.
* Other experimental drugs are being used.
* Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | 1 year after treatment completion
  complete response (CR) rate, evaluated by PET-CT and CT/MRI, according to Lugano 2014 criteria

SECONDARY OUTCOMES:
overall response rate (ORR) | 1 year after treatment completion
  overall response rate (ORR), evaluated by PET-CT and MRI, according to Lugano 2014 criteria
1-year progression free survival rate (PFS) | 1 year after treatment completion
  1-year progression free survival rate (PFS), time from date of enrolment to date of disease progression, death of any reason, whichever comes first
1-year overall survival rate (OS) | 1 year after treatment completion
  1-year overall survival rate (OS), time from date of enrolment to date of death of any reason.
adverse events according to CTCAE 5.0 | 1 year after treatment completion
  safety profiles, evaluated by adverse events according to CTCAE 5.0
disease control rate (DCR) | 1 year after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, Ph.D, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feng Y, Rao H, Lei Y, Huang Y, Wang F, Zhang Y, Xi S, Wu Q, Shao J. CD30 expression in extranodal natural killer/T-cell lymphoma, nasal type among 622 cases of mature T-cell and natural killer-cell lymphoma at a single institution in South China. Chin J Cancer. 2017 May 10;36(1):43. doi: 10.1186/s40880-017-0212-9. PMID 28486951
- [Result] Kwong YL, Kim WS, Lim ST, Kim SJ, Tang T, Tse E, Leung AY, Chim CS. SMILE for natural killer/T-cell lymphoma: analysis of safety and efficacy from the Asia Lymphoma Study Group. Blood. 2012 Oct 11;120(15):2973-80. doi: 10.1182/blood-2012-05-431460. Epub 2012 Aug 23. PMID 22919026
- [Result] Kwong YL, Chan TSY, Tan D, Kim SJ, Poon LM, Mow B, Khong PL, Loong F, Au-Yeung R, Iqbal J, Phipps C, Tse E. PD1 blockade with pembrolizumab is highly effective in relapsed or refractory NK/T-cell lymphoma failing l-asparaginase. Blood. 2017 Apr 27;129(17):2437-2442. doi: 10.1182/blood-2016-12-756841. Epub 2017 Feb 10. PMID 28188133
- [Result] Li X, Cheng Y, Zhang M, Yan J, Li L, Fu X, Zhang X, Chang Y, Sun Z, Yu H, Zhang L, Wang X, Wu J, Li Z, Nan F, Tian L, Li W, Young KH. Activity of pembrolizumab in relapsed/refractory NK/T-cell lymphoma. J Hematol Oncol. 2018 Jan 31;11(1):15. doi: 10.1186/s13045-018-0559-7. PMID 29386072
- [Result] Chan TSY, Li J, Loong F, Khong PL, Tse E, Kwong YL. PD1 blockade with low-dose nivolumab in NK/T cell lymphoma failing L-asparaginase: efficacy and safety. Ann Hematol. 2018 Jan;97(1):193-196. doi: 10.1007/s00277-017-3127-2. Epub 2017 Sep 6. No abstract available. PMID 28879531
- [Result] Tao R, Fan L, Song Y, Hu Y, Zhang W, Wang Y, Xu W, Li J. Sintilimab for relapsed/refractory extranodal NK/T cell lymphoma: a multicenter, single-arm, phase 2 trial (ORIENT-4). Signal Transduct Target Ther. 2021 Oct 27;6(1):365. doi: 10.1038/s41392-021-00768-0. PMID 34702811
- [Result] Kim HK, Moon SM, Moon JH, Park JE, Byeon S, Kim WS. Complete remission in CD30-positive refractory extranodal NK/T-cell lymphoma with brentuximab vedotin. Blood Res. 2015 Dec;50(4):254-6. doi: 10.5045/br.2015.50.4.254. Epub 2015 Dec 21. No abstract available. PMID 26770954
- [Result] Advani RH, Moskowitz AJ, Bartlett NL, Vose JM, Ramchandren R, Feldman TA, LaCasce AS, Christian BA, Ansell SM, Moskowitz CH, Brown L, Zhang C, Taft D, Ansari S, Sacchi M, Ho L, Herrera AF. Brentuximab vedotin in combination with nivolumab in relapsed or refractory Hodgkin lymphoma: 3-year study results. Blood. 2021 Aug 12;138(6):427-438. doi: 10.1182/blood.2020009178. PMID 33827139
- [Result] Yamaguchi M, Suzuki R, Oguchi M, Asano N, Amaki J, Akiba T, Maeda T, Itasaka S, Kubota N, Saito Y, Kobayashi Y, Itami J, Ueda K, Miyazaki K, Ii N, Tomita N, Sekiguchi N, Takizawa J, Saito B, Murayama T, Ando T, Wada H, Hyo R, Ejima Y, Hasegawa M, Katayama N. Treatments and Outcomes of Patients With Extranodal Natural Killer/T-Cell Lymphoma Diagnosed Between 2000 and 2013: A Cooperative Study in Japan. J Clin Oncol. 2017 Jan;35(1):32-39. doi: 10.1200/JCO.2016.68.1619. Epub 2016 Oct 31. PMID 28034070
- [Result] Lim SH, Hong JY, Lim ST, Hong H, Arnoud J, Zhao W, Yoon DH, Tang T, Cho J, Park S, Ko YH, Kim SJ, Suh C, Lin T, Kim WS. Beyond first-line non-anthracycline-based chemotherapy for extranodal NK/T-cell lymphoma: clinical outcome and current perspectives on salvage therapy for patients after first relapse and progression of disease. Ann Oncol. 2017 Sep 1;28(9):2199-2205. doi: 10.1093/annonc/mdx316. PMID 28911074